CLINICAL TRIAL: NCT01747499
Title: Phase I/II Trial of Intravenous Azacitidine in Patients Undergoing Matched Unrelated Stem Cell Transplantation
Brief Title: Azacitidine in Patients Undergoing Matched Unrelated Stem Cell Transplantation
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Enrolling 8 more patients would be statistically unlikely that the primary endpoint would be reached (reduce day 180 grade II-IV GVHD rates to 20% or less)
Sponsor: Washington University School of Medicine (Other)
Collaborators: The Foundation for Barnes-Jewish Hospital (Other); National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201303012; 1P50CA171963-01A1 (NIH)
Record Dates: First submitted 2012-12-07; First posted 2012-12-11 (Estimated); Results first posted 2019-10-16 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-09

CONDITIONS: Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Precursor Cell Lymphoblastic Leukemia-Lymphoma
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): Conditioning treatment
  Transplant on Day 0
  15 mg/m^2 azacitidine Days 7-11
  15 mg/m^2 azacitidine Days 35-39
  15 mg/m^2 azacitidine Days 63-67
  15 mg/m^2 azacitidine Days 91-95
  Interventions: Drug: Azacitidine
- Cohort 2 (Experimental): Conditioning treatment
  Transplant on Day 0
  30 mg/m^2 azacitidine Days 7-11
  30 mg/m^2 azacitidine Days 35-39
  30 mg/m^2 azacitidine Days 63-67
  30 mg/m^2 azacitidine Days 91-95
  Interventions: Drug: Azacitidine
- Cohort 3 (Experimental): Conditioning treatment
  Transplant on Day 0
  37.5 mg/m^2 azacitidine Days 7-11
  37.5 mg/m^2 azacitidine Days 35-39
  37.5 mg/m^2 azacitidine Days 63-67
  37.5 mg/m^2 azacitidine Days 91-95
  Interventions: Drug: Azacitidine
- Cohort 4 (Experimental): Conditioning treatment
  Transplant on Day 0
  45 mg/m^2 azacitidine Days 7-11
  45 mg/m^2 azacitidine Days 35-39
  45 mg/m^2 azacitidine Days 63-67
  45 mg/m^2 azacitidine Days 91-95
  Interventions: Drug: Azacitidine
- Phase II Cohort (Experimental): Conditioning treatment
  Transplant on Day 0
  Dose determined in Phase I - 45 mg/m^2 azacitidine Days 7-11
  Dose determined in Phase I - 45 mg/m^2 azacitidine Days 35-39
  Dose determined in Phase I - 45 mg/m^2 azacitidine Days 63-67
  Dose determined in Phase I - 45 mg/m^2 attitudinize Days 91-95
  Interventions: Drug: Azacitidine

INTERVENTIONS:
Drug: Azacitidine
  Other Names: Vidaza®; Ladakamycin; 5-AzaC

SUMMARY:
The purpose of this phase I/II study is to define the maximum tolerated dose of 5-AzaC and the effect on grade II-IV GvHD when given after matched unrelated donor transplant (MUD).

ELIGIBILITY:
Inclusion Criteria:

Patients must meet the following criteria within 30 days prior to Day 0 unless otherwise noted.

* Phase I: Diagnosis of any hematological malignancy listed below (excluding myelofibrosis) in remission or with stable minimal residual disease

  * Acute myelogenous leukemia (AML) in 1st or subsequent remission or in relapse after any remission
  * Acute lymphoblastic leukemia (ALL) in 1st or subsequent remission or in relapse after any remission
  * Myelodysplastic syndrome either intermediate 1 or 2, or high risk by the International Prognostic Scoring System
  * Chronic myelogenous leukemia (CML) in accelerated or second chronic phase
  * Non-Hodgkin's lymphoma (NHL) or Hodgkin's disease (HD) in 2nd or greater complete remission, partial remission, or refractory relapse
  * Chronic lymphocytic leukemia (CLL), Rai Stage 2-4, failing at least 2 prior regimens
  * Multiple myeloma (MM), Stage 2-3
  * Myeloproliferative disorder or neoplasm
* Phase II: Diagnosis of AML in remission 1 or 2 or a diagnosis of myelodysplastic syndrome either intermediate 1 or 2, or high risk by the International Prognostic Scoring System.
* Patients with MDS must be transplant candidates by current clinical standards.
* Patients who have been treated with hypomethylating agents prior to entering the study are eligible.
* Must have matched unrelated donor (8 of 8 HLA match at A, B, C, and DR loci) by high resolution DNA typing
* Must have donor peripheral blood stem cells mobilized by NMDP standards. No bone marrow donors.
* Must have 2-8 x 10^6 CD34+ cells/kg (recipient weight) infused on Day 0.
* Must have at least one additional aliquot of >=1 x 10^6 CD34/kg cryopreserved cells stored at the time of transplant.
* Must receive a myeloablative or reduced intensity conditioning regimen for SCT as defined by the CIBMTR

  * Cyclophosphamide and single dose total body irradiation
  * Fludarabine and busulfan
  * Fractionated TBI and cyclophosphamide
  * Busulfan and cyclophosphamide
* Must be able to receive GVHD prophylaxis with tacrolimus and methotrexate.
* Must be ≥ 18 yrs old and ≤ 70 yrs old. Azacitidine is not approved by the FDA for use in children.
* Must have an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* Must have laboratory results indicating:

  * Total bilirubin < 2.0 mg/dl, unless a diagnosis of Gilbert's disease
  * AST/ALT ≤ 3 X the upper limit of institutional normal
  * Serum creatinine ≤ 2.0 mg/dl
* Patient must have ability to understand and willingness to provide written informed consent prior to participation in the study and any related procedures being performed.
* The effects of azacitidine on the developing human fetus at the recommended therapeutic dose are unknown. For this reason and because category D agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of childbearing age must have a negative serum pregnancy test (ß-human chorionic gonadotropin) within 72 hours prior to initiating the conditioning regimen and be willing to not become pregnant by using effective contraception while undergoing treatment and for at least 3 months after the last dose of azacitidine.
* Men must be willing not to father a new child while receiving therapy. They must use an effective barrier method of contraception during the study and for 3 months following the last dose.

Exclusion Criteria:

* Must not have myelofibrosis or other disease known to prolong neutrophil engraftment to > 28 days after transplant.
* Must not be receiving any other investigational agents within 14 days of first dose of azacitidine (Day 7).
* Must not have myeloablative conditioning as defined below:

  * TBI < or = Gy +/- purine analog
  * Flu + Cy +/- ATG
  * Flu + AraC + Ida
  * Cladribine + AraC
  * Total Lymphoid Irradiation + ATG
* Must not receive antithymocyte globulin as part of pre-transplant conditioning regimens. Antithymocyte globulin is excluded due to its potential impact on modulating the incidence of GvHD or GvL.
* Must not have uncontrolled intercurrent illness including ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements.
* Must not be pregnant or breastfeeding. Pregnant women are excluded from this study because azacitidine is a Category D agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with azacitidine, breastfeeding should be discontinued if the mother is treated azacitidine. These potential risks may also apply to other agents used in this study.
* Must not have a known or suspected hypersensitivity to azacitidine, mannitol, or compounds of similar composition to azacitidine..
* Must not have an advanced malignant hepatic tumor.
* Must not be HIV, HBV, or HCV positive.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2013-04-15; Primary Completion 2018-08-31 (Actual); Study Completion 2018-12-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark A. Schroeder, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Phase II Cohort
Started | 3 | 3 | 3 | 6 | 39
Completed | 2 | 2 | 3 | 4 | 24
Not Completed | 1 | 1 | 0 | 2 | 15
Not completed — Steroid refractory aGvHD | 1 | 0 | 0 | 1 | 4
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 2
Not completed — Death | 0 | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 6
Not completed — Developed AML and death | 0 | 0 | 0 | 0 | 1
Not completed — Determined not to be eligible | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Phase II Cohort | Total
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 39 | 54
Age, Continuous [Median (Full Range); unit: years] | 46 [27 to 56] | 57 [51 to 63] | 63 [39 to 63] | 58.5 [36 to 69] | 59 [24 to 70] | 59 [24 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 0 | 2 | 17 | 22
  Male | 2 | 1 | 3 | 4 | 22 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 3 | 6 | 39 | 54
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 1 | 1
  White | 3 | 3 | 3 | 5 | 37 | 51
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 6 | 39 | 54

OUTCOME MEASURES:

1. Primary Outcome: Phase I: to Determine the Maximum Tolerated Dose (MTD) of Azacitidine in Patients Undergoing Matched (8 Out of 8) Unrelated Donor Transplant for Any Hematological Malignancy in Remission or With Stable Disease.
Description: The MTD is defined as the dose level immediately below the dose level at which patients of a cohort (of 2 to 6 patients) experience dose-limiting toxicity.
Time Frame: 28 days
Measure: Number; unit: mg/m^2
Groups:
- Phase I: Conditioning treatment
  Transplant on Day 0
  Azacitidine Days 7-11
  Azacitidine Days 35-39
  Azacitidine Days 63-67
  Azacitidine Days 91-95
Arm/Group | Phase I
Number analyzed (Participants) | 15
mg/m^2 | 45

2. Primary Outcome: Phase II: Number of Participants With Grades II-IV Acute GvHD
Description: GVHD rate and severity will be assessed based on modified Glucksberg criteria. Grade II-IV and III-IV aGVHD in first 180 days after transplant will be assessed.
Time Frame: Day +180
Population: One patient was enrolled and treated with 1 cycle but was ultimately ineligible following a laboratory error and is not evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II Cohort
Number analyzed (Participants) | 38
Participants | 16

3. Secondary Outcome: Rate of Grades III-IV aGVHD at Day +180.
Description: GVHD rate and severity will be assessed based on modified Glucksberg criteria.
Time Frame: Day +180
Population: One patient in Phase II cohort was enrolled and treated with 1 cycle but was ultimately ineligible following a laboratory error and is not evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Phase II Cohort
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 38
Participants | 0 | 0 | 0 | 0 | 9

4. Secondary Outcome: Overall Survival as Measured by Number of Participants Alive at 1 Year After Transplant
Description: Date of transplant to the date of death from any cause.
Time Frame: One year after transplant
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Phase II Cohort
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 38
Participants | 3 | 2 | 2 | 4 | 28

5. Secondary Outcome: Treatment-related Mortality
Description: Death that results from a transplant procedure-related complication (e.g. infection, organ failure, hemorrhage, GVHD) rather than from relapse of the underlying disease or an unrelated cause.
Time Frame: Day +140
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Phase II Cohort
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 38
Participants | 0 | 0 | 0 | 1 | 2

6. Secondary Outcome: Number of Participants Who Relapsed Within the First Year of Transplant
Description: Recurrence of the original malignant disease after transplantation. The time to relapse is the time to the first observation of hematologic, radiographic, or cytogenetic changes, which result in characterization as relapse.
Time Frame: Within the first year of transplant
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Phase II Cohort
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 38
Participants | 1 | 0 | 1 | 1 | 4

7. Secondary Outcome: Rate of Chronic GvHD
Time Frame: One year after transplant
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Phase II Cohort
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 38
Participants | 3 | 2 | 2 | 3 | 27

ADVERSE EVENTS:
Time Frame: -Adverse events (AEs) were collected from Day +7-Day +140 visit or 30 days after their last dose of azacitidine (for patients that did not complete all 4 cycles of treatment). -All AEs were collected for Phase I patients -Only selected adverse events were collected for Phase II patients *all grade 3, 4, or 5 *any that require azacitidine treatment to be delayed, held, or discontinued *any that require modification of GVHD prophylaxis medications *any grade mucositis and any infection
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Phase II Cohort
All-Cause Mortality (participants affected / at risk) | 1/3 | 1/3 | 1/3 | 2/6 | 12/39
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/3 | 2/3 | 3/6 | 23/39
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 6/6 | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=3) | Cohort 3 (N=3) | Cohort 4 (N=6) | Phase II Cohort (N=39)
Fever (General disorders) | 1 | 0 | 0 | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Hypoxic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Relapsed acute leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Acute kidney failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 6
Sepsis (Infections and infestations) | 0 | 0 | 0 | 3 | 1
Hematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Vascular access complication (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pruritic rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 5
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Respiratory infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
HHV-6 (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Edema limbs (General disorders) | 0 | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=3) | Cohort 3 (N=3) | Cohort 4 (N=6) | Phase II Cohort (N=39)
Anemia (Blood and lymphatic system disorders) | 2 | 1 | 1 | 5 | 14
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 2 | 5
Hemolysis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1
Hemolytic uremic syndrome (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 1 | 2
Heart failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 2
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 1 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Tachycardia (NOS) (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cushingoid (Endocrine disorders) | 0 | 0 | 0 | 2 | 0
Dry eye (Eye disorders) | 1 | 0 | 0 | 0 | 0
Vision changes (not otherwise specified) (Eye disorders) | 0 | 0 | 0 | 1 | 0
Watering eyes (Eye disorders) | 1 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Bloating (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 1 | 2 | 3 | 4
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 1
Mouth gumminess (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 3 | 1 | 1 | 6 | 20
Nausea (Gastrointestinal disorders) | 3 | 2 | 2 | 2 | 0
Oral hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Sore in mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 2 | 1 | 3 | 0
Chills (General disorders) | 2 | 1 | 0 | 1 | 0
Edema limbs (General disorders) | 2 | 1 | 0 | 3 | 2
Fatigue (General disorders) | 1 | 0 | 1 | 1 | 4
Fever (General disorders) | 0 | 1 | 0 | 1 | 0
Flu Like Symptoms (General disorders) | 0 | 0 | 0 | 1 | 0
Localized edema (General disorders) | 1 | 0 | 0 | 0 | 0
Neck edema (General disorders) | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 3
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Allergic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 1
BK virus (Infections and infestations) | 0 | 0 | 0 | 0 | 1
C. Difficile (Infections and infestations) | 0 | 0 | 0 | 0 | 2
CMV Positive Culture (Infections and infestations) | 2 | 0 | 0 | 0 | 0
CMV Viremia (Infections and infestations) | 1 | 1 | 1 | 0 | 3
Catheter related infection (Infections and infestations) | 1 | 1 | 0 | 0 | 1
Coagulase Negative Staphyloccus-Bacteremia (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Coronavirus OC43 Parainfluenza virus Type 3 (Infections and infestations) | 0 | 0 | 0 | 0 | 1
E. coli bacteremia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Healthcare associated pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Hepatic infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Influenza A (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 0 | 1 | 2
Mucosal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 4
Papulopustular rash (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Rhinovirus positive culture (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Sinusitis (rhinovirus/enterovirus) (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0 | 1 | 1
Streptococcus mitis bacteremia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Upper respiratory infection (Infections and infestations) | 0 | 1 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 3
Bruising (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Dog bite to finger (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 0 | 3 | 2
Alanine aminotransferase increased (Investigations) | 2 | 2 | 3 | 4 | 6
Alkaline phosphatase increased (Investigations) | 0 | 2 | 2 | 4 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 3 | 4 | 2
Blood bilirubin increased (Investigations) | 1 | 1 | 0 | 3 | 4
Creatinine increased (Investigations) | 0 | 1 | 2 | 3 | 2
Ejection fracture decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Fibrinogen decreased (Investigations) | 0 | 0 | 0 | 0 | 1
INR increased (Investigations) | 1 | 3 | 0 | 5 | 0
Lymphocyte count decreased (Investigations) | 2 | 1 | 0 | 4 | 17
Neutrophil count decreased (Investigations) | 2 | 0 | 0 | 3 | 21
Platelet count decreased (Investigations) | 2 | 2 | 1 | 5 | 20
Weight loss (Investigations) | 0 | 0 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 2 | 1 | 1 | 5 | 15
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 2 | 5
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 3 | 12
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 2 | 3 | 5 | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 1
Hypernatremia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 2 | 0 | 2 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 5 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 3 | 0 | 2 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 4 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 1 | 3 | 4 | 0
Hyponatremia (Metabolism and nutrition disorders) | 2 | 2 | 3 | 6 | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 3 | 1 | 1 | 5 | 14
Iron overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 2 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 3
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 2 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Drooling (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Facial droop (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Facial muscle weakness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 1 | 0 | 2 | 0
Hypersomnia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Paresthesia (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Sinus pain (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Stroke (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Altered mental status (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0
Confusion (Psychiatric disorders) | 0 | 2 | 1 | 2 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0
Hallucinations (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 2 | 1 | 3 | 3
Bladder spasm (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Hematuria (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 2
Proteinuria (Renal and urinary disorders) | 1 | 1 | 0 | 1 | 0
Urinary frequency (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Perianal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Acute worsening of COPD (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 0
Blanching erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Erythema (face) (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0
Erythema at catheter site (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Lip ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 2
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Rash (sun burn) (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 5 | 10
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 2 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Hot flashes (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 4
Hypotension (Vascular disorders) | 1 | 1 | 0 | 2 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Thromboembolic event (Vascular disorders) | 0 | 0 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-06): https://cdn.clinicaltrials.gov/large-docs/99/NCT01747499/Prot_SAP_000.pdf